CLINICAL TRIAL: NCT01506921
Title: A Prospective Randomised, Double-blinded Cross-over Study to Investigate the Effects of Racemic and S-ketamine on Cerebral Blood Flow on Healthy Volunteers With MRI-ASL
Brief Title: Racemic Ketamine Versus S-ketamine With Arterial Spin Labeling (ASL)-MRI in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Anders Schmidt, principal investigator, Lund University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 11 MRI-ASL
Record Dates: First submitted 2011-12-28; First posted 2012-01-10 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Healthy; Abnormal Vascular Flow
Keywords: racemic ketamine; S-ketamine; Cerebral blood flow; Magnetic resonance imaging; arterial spin labeling; healthy volunteers
MeSH Terms: interventions — Ketamine; Esketamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Racemic ketamine (Active Comparator)
  Interventions: Drug: Racemic ketamine
- S-ketamine (Active Comparator): All subjects receive both study drugs in a cross- over design. Equipotent doses are used. 0,6 mg/kg racemic ketamine equals 0,3 mg/kg s-ketamine
  Interventions: Drug: S-ketamine

INTERVENTIONS:
Drug: Racemic ketamine — 0.6 mg/kg
  Other Names: Ketamine
  Arms: Racemic ketamine
Drug: S-ketamine — 0.3 mg/kg
  Other Names: Ketanest
  Arms: S-ketamine

SUMMARY:
Racemic ketamine and S-ketamine are used in clinical practice today. Little is known of their difference in effect on cerebral blood flow, volume and metabolism. cerebral blood flow (CBF) measuring techniques are limited in time so constant measurement to mirror a dynamic process is impossible or very difficult. A novel MRI application, arterial spin labeling, offers the possibility that without radiation or contrast, to measure semi-continuous CBF with measurements every 60-120 seconds. The investigators will give 14 healthy volunteers both study drugs in a randomised sequence with one week apart and measure regional CBF during the study period of 45 minutes after a sub-anaesthetic bolus dose of 0,6 mg/kg racemic ketamine and 0,3 mg/kg S-ketamine The investigators hypothesize that there is no difference between racemic ketamine and S(+)-ketamine with regards to Arterial Spin Labeling (ASL) measured cerebral blood flow.

DETAILED DESCRIPTION:
In this investigator-initiated randomised, double-blinded, crossover study, adult healthy volunteers will be randomised to receive, as 60-second iv bolus injections on two different occasions with at least seven days interval, 0.3 mg kg of S-ketamine (Ketanest® 5.0 mg/ ml, Pfizer, USA) or 0.6 mg/kg of racemic ketamine (Ketalar® 10 mg/ml, Pfizer, USA) supplied by the hospital pharmacy.

The volunteers will consecutively be given specific inclusion numbers and randomized according to a schedule with corresponding randomization codes prepared in advance by the Research & Development Centre of the Skåne Region, Skåne University Hospital, Lund, Sweden. Before each investigation, a sealed envelope marked with the corresponding inclusion number, will be opened in a separate room by a nurse not taking further part in the study. The nurse prepared the study drug according to the randomization code in a 20 ml syringe based on a bodyweight-based dosing schedule, and diluted the study drug with saline to a total volume of 20 ml. The prepared syringe, marked with the inclusion number, date and signature, will be handed over to the investigator.

After an initial 10-minute period of dynamic baseline measurements, the study drug will be injected manually by the investigator. ASL measurements will be made over a 45-minute study period starting from the injection of study drug, and the volunteer will be brought to the preparation room for at least 60 minutes of further supervision until clinical routine criteria for postoperative discharge will be met.

Fourteen healthy (American Society of Anaesthesiologists physical status 1) adult volunteers will be included after physical examinations and individual written informed consents. Female subjects will be required to use effective anti-conception methods during the study period. The volunteers will have to refrain from caffeine, nicotine, alcohol and medications for 72 hours, and fast for six hours, but will be allowed to drink water until two hours before each ASL-MRI investigation.

Each volunteer will be offered ear plugs, asked to rest with eyes closed during the scanning procedure, and left undisturbed throughout the study period. Oxygen 2 l/min will be delivered by nasal cannula.

A hand vein will be cannulated with a 20 G (1.1 mm) 45 mm teflon catheter for injection of study drug, and a balanced glucose solution will be infused at a rate of 1.0 ml/kg/h iv. The radial artery will be cannulated at wrist level with a 20 G 45 mm teflon catheter after local infiltration with 2-3 ml of lidocaine. Each volunteer will be connected to an N-MRI2-01 monitoring device recording the ECG, invasive blood pressure, SpO2, ETCO2 and respiratory rate.

Monitored data will be sampled minutely throughout the study period, saved onto a PC card and analyzed with the Datex-Ohmeda S/5Collect version 4.0™ software package.

Arterial blood for blood gas analysis was obtained at baseline and at 1, 5, 10 and 15 min after injection of the study drug. Analyses were made on a Radiometer ABL800 FLEX device The ASL data will be acquired using a 3 Tesla MRI unit. A three-dimensional (3D) GRASE pulse sequence will be employed (2), using a labeling and saturation schedule based on FAIR (3) and Q2TIPS (4).

Drug-induced changes in regional perfusion will be monitored over time using a single inversion time (TI) of 2000 ms and repeated 115 times, and a repetition time (TR) of 3000 ms. For multiple TI, ten time points were acquired with a starting point at TI = 300 ms and an increment of 300 ms between time points, the total inflow time was 1400 ms and the TR was set to 3700 ms.

Data sets will be preprocessed using realign tools of the Statistical Parameters Mapping version 8.0 (SPM8) software package (Wellcome Department of Imaging Neuroscience, London, UK; http://www.fil.ion.ucl.ac.uk/spm) and executed in the Matlab 7.11 software package. The labeled and control images will be pair-wise subtracted to produce CBF-weighted ASL images from re-aligned control/tag images, and these difference maps were denoised using an established wavelet-domain filtering method (5), and an in-house software program written in IDL 7.1 (ITT Visual Information Solutions, Boulder, CO, USA). Values of CBF (in ml/100g/min) will be calculated using a general kinetic model (6) according to the Buxton equation CBF values will be determined by drawing different numbers of symmetrical cerebral regions of interest (ROI) bilaterally to outline the grey matter of the frontal lobes, parietal lobes, temporal lobes, occipital lobes, insular cortex, anterior cingulate, posterior cingulate, thalamus, caudate nucleus and putamen. Global CBF values will determined by drawing a large ROI to outline the whole brain tissue within the skull.

ELIGIBILITY:
Inclusion Criteria:

* healthy (ASA 1),
* age 18-65 years,
* fertile women must use approved anticonception during study period (2 weeks)

Exclusion Criteria:

* known or suspected pregnancy,
* BMI < 30,
* motion sickness,
* claustrophobia,
* somatic or psychiatric disease,
* drug abuse,
* chronic medication,
* drug allergy,
* difficulties in understanding the written and spoken Swedish language

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2011-05; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
regional cerebral blood flow | - Measured every 30 seconds from baseline to 45 min after study drug injection
  -In ml/100g/min

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Åkeson, profesor, Study Director — Lund University
Locations (1):
- Deprtment of radiology, SUS, Malmö, Malmo, Malmö, Sweden